CLINICAL TRIAL: NCT01022931
Title: Evaluation of a New Virus(Influenza A H1N1/09) in Children: Epidemiology, Clinical Presentation and Outcome, and Response to Treatment
Brief Title: Epidemiology and Clinical Presentation of H1N1 Infection in Children in Geneva
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Klara M. Pósfay Barbe, Head of Pediatric Infectious Diseases, University Hospital, Geneva
Other Study IDs: H1N1epidemiology
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Healthy; Immunosuppressed; Asthmatic; Neuromuscular Diseases
Keywords: Influenza A H1N1; Children; Epidemiology; Treatment; Oseltamivir; Genetics
MeSH Terms: conditions — Asthma; Neuromuscular Diseases; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swab; DNA for genetic polymorphisms (Response to oseltamivir)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to identify clinical symptoms and outcomes, as well as response to anti-viral treatment in children living in Geneva, with influenza A/ H1N1 infection during the current pandemic.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of H1N1 infection

Exclusion Criteria:

* Not available for a 30 days follow-up

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children seen at the emergency ward
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
ABCB1 polymorphisms | 6 months
  ABCB1 gene polymorphisms and neuropsychiatric adverse events in oseltamivir-treated children during influenza H1N1/09 pandemia

CONTACTS AND LOCATIONS:
Overall Officials: Klara M Posfay-Barbe, MD, MS, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Children's Hospital of Geneva, HUG, Geneva, Canton of Geneva, Switzerland